CLINICAL TRIAL: NCT04490720
Title: The Efficacy Evaluation of Buckwheat Husk Extract on Cardiovascular Disease Risk Factors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201911003RSC
Record Dates: First submitted 2020-07-26; First posted 2020-07-29 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): consume 1 sachet per day for 2 months
  Interventions: Dietary Supplement: Placebo
- Buckwheat husk extract (Experimental): consume 1 sachet per day for 2 months
  Interventions: Dietary Supplement: Buckwheat husk extract

INTERVENTIONS:
Dietary Supplement: Placebo — consume 1 sachet per day for 2 months
  Arms: Placebo
Dietary Supplement: Buckwheat husk extract — consume 1 sachet per day for 2 months
  Arms: Buckwheat husk extract

SUMMARY:
To assess the efficacy evaluation of buckwheat husk extract on cardiovascular disease risk factors

DETAILED DESCRIPTION:
This is a double-blind and randomized study. Subjects are informed to consume the samples every day for 2 months. The clinical diagnosis item of cardiovascular disease is evaluated by the doctor.

ELIGIBILITY:
Inclusion Criteria:

1. 20 to 65-year-old males or non-pregnant females who are willing to sign the subject's consent.
2. The systolic blood pressure is 121-139 mmHg and the diastolic blood pressure is between 81-89 mmHg.
3. Those who are not pregnant and are willing to cooperate with contraception during the trial period.
4. No history of organ transplantation, epilepsy or convulsions, liver or kidney disease, malignant tumor, endocrine disease, mental disease, alcohol or drug abuse, or other major organic diseases (according to medical history).

Exclusion Criteria:

1. Pregnant women.
2. People with a history of organ transplantation, epilepsy or convulsions, liver and kidney disease, malignant tumors, endocrine diseases, mental illness, alcohol or drug abuse, and other major organic diseases (according to medical history).
3. No person has undergone major surgery.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in blood pressure (systolic blood pressure, diastolic blood pressure) | Days 1, 28, and 56
  Blood pressure will be measured at the beginning, 4-week, and 8-week time points.

SECONDARY OUTCOMES:
Change from baseline in Body Mass Index (BMI) | Days 1, 28, and 56
  Body Mass Index (kg/m^2) will be measured at the beginning, 4-week, and 8-week time points.
  P.S. weight in kilograms, height in meters
Change from baseline in waist-hip ratio | Days 1, 28, and 56
  Waist-hip ratio will be measured at the beginning, 4-week, and 8-week time points.
Change from baseline in blood lipid (total-Cholesterol, triglyceride, HDL-C, LDL-C) | Days 1, 28, and 56
  Blood lipid will be measured at the beginning, 4-week, and 8-week time points.
Change from baseline in blood cardiovascular disease risk biomarker (hs-CRP, NO, Trimethylamine-N-oxide) | Days 1, 28, and 56
  Blood cardiovascular disease risk biomarker will be measured at the beginning, 4-week, and 8-week time points.

CONTACTS AND LOCATIONS:
Overall Officials: Mao-Hsin Lin, Doctor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan